CLINICAL TRIAL: NCT05960513
Title: Impact of Breathing Exercises and Meditation on Improving Quality of Life in Glaucoma Patients: An Electronic Pilot Feasibility Study
Brief Title: Impact of Breathing Exercises and Meditation on Improving Quality of Life in Glaucoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Monali Malvankar, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 122096
Record Dates: First submitted 2023-07-14; First posted 2023-07-25 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Glaucoma; Depression; Anxiety; Quality of Life; Sleep Disorder
Keywords: Health-related Quality of Life; Glaucoma; COVID-19; Breathing; Meditation
MeSH Terms: conditions — Glaucoma; Depression; Anxiety Disorders; Sleep Wake Disorders; COVID-19; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercises followed by Meditation (Experimental): Breathing exercises and Meditation taught by Prasanna Wellness, a non-profit organization, helps dissolve stress and create a proper system in the mind. These breathing exercises include slow deep breaths and rapid breaths and are followed by meditation. Participants will receive three weekly online instructions (90 minutes each) by trained instructors in addition to standard care. Weekly 60 minutes follow-ups will include 10 minutes of breathing exercises followed by 33 minutes of guided meditation practice, and then focus on participants' experiences with breathing exercise followed by meditation during the week, additional observations, and a review of relevant knowledge to support their home practice.
  Interventions: Behavioral: Breathing Exercises followed by Meditation
- No Intervention (No Intervention): The usual standard of care for patients with glaucoma includes starting them on first line of drugs. Participants will be initiated and maintained on appropriate dosages of such medications as part of standard of care. The usual standard of care also includes an ophthalmic examination measuring best-corrected Snellen VA and pinhole acuities and a follow-up visit once a year.

INTERVENTIONS:
Behavioral: Breathing Exercises followed by Meditation — Breathing exercises and Meditation taught by Prasanna Wellness, a non-profit organization, helps dissolve stress and create a proper system in the mind. These breathing exercises include slow deep breaths and rapid breaths and are followed by meditation. Meditation is a guided meditation that helps to eliminate stress and establish an apposite system in the mind, therefore inducing physiological and mental relaxation whilst the eyes are shut. The proposed duration and frequency of the follow-up will be 60-minutes weekly for 11 weeks.
  Arms: Breathing Exercises followed by Meditation

SUMMARY:
Glaucoma is a chronic disease that causes loss of vision and potentially blindness as a result of optic nerve damage, often due to increased intraocular pressure. Glaucoma is currently the leading cause of irreversible blindness worldwide.1 In 2020, 4.1 million and 3.6 million adults over the age of 50 suffered from mild to severe glaucoma-induced visual impairment and blindness, respectively.1 However, these figures are likely underestimated since glaucoma can remain asymptomatic until later stages in disease progression.2 The relaxation response evoked by mind-body interventions, such as breathing exercises and meditation, is known to reduce stress and improve quality of life (QOL). In a recent study, mindfulness-based meditation was found to reduce intraocular pressure and improve QOL in patients with glaucoma.3 A feasibility study will be conducted using a mixed-method design to assess the feasibility of the online delivery of an intervention titled Breathing Exercises followed by Meditation for potentially enhancing the QOL and mental health of glaucoma patients. Upon recruitment, participants will undergo blocked randomization to either the intervention arm or usual care arm, stratified by sex. Participants in each arm will complete online questionnaires at baseline and after 12 weeks to collect data on health-related quality of life (HRQOL), depression symptoms, anxiety, and sleep quality using REDCap, an electronic data capturing system provided by Lawson Health Research Institute (LHRI). Our study can help to assess the feasibility of conducting a pilot study on breathing exercises followed by meditation to assess its effects in a sample of patients with glaucoma.

ELIGIBILITY:
Inclusion and Exclusion Criteria Inclusion Criteria

1. Patients diagnosed with glaucoma.
2. Patients aged 40-65.
3. Being able to provide valid informed consent to participate in the research study.
4. Being able to read and understand English.
5. Having no significant self-reported or physician-diagnosed mental health disorder.
6. Independent access to a computer to participate in virtual sessions.
7. Must be able to sit comfortably for 30-35 minutes without any major pain or discomfort, can hear well enough to follow verbal instructions when the eyes are closed, and be in good general physical health.

Exclusion Criteria

1. Inability to provide valid informed consent.
2. Significant communication barriers or lack of English proficiency that prevents participants from completing the questionnaires.
3. Severe depression as confirmed by a CES-D ≥ 24.
4. Having a lifetime diagnosis of self-reported other serious mental disorders, including bipolar I or II disorder, primary psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder).
5. Self-reported substance abuse or dependence within the past 3 months.
6. Having acutely unstable medical illnesses, including delirium or acute cerebrovascular or cardiovascular events within the last 6 months.
7. Having irreversible vision loss that prevents one from completing the questionnaires.
8. Participation in a study involving similar techniques.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life (HRQoL) | Baseline visit, Week 1, Week 3, Week 6, Week 12
  HRQoL is an essential measure of quality of life related to health; it helps physician identify hidden morbidity in clinical care as well as improves patient-physician communications. HRQoL will be measured using time trade-off questionnaire
Change in Depression | Baseline visit, Week 1, Week 3, Week 6, Week 12
  Depression is a feeling of severe despondency and dejection. Depression will be measured using the Center for Epidemiological Studies - Depression (CES-D) score.
Change in Anxiety | Baseline visit, Week 1, Week 3, Week 6, Week 12
  Anxiety will be measured using Hospital Anxiety and Depression Scale - Anxiety (HADS-A) subscale
Change in Sleep quality | Baseline visit, Week 1, Week 3, Week 6, Week 12
  Sleep quality as measured using the Pittsburgh Sleep Quality Index (PSQI) scores.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital, Ivey Eye Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) collected in this study will not be available to other researchers (e.g., outside the primary research group). Since the primary research group has the necessary expertise to analyze the data and do not need any outside help.